CLINICAL TRIAL: NCT03463512
Title: Multicenter, Open-label, Controlled, Randomized Clinical Study to Evaluate the Efficacy and Safety of Racecadotril in Infants, Children and Adolescents With Acute Diarrhea
Brief Title: Controlled Study to Evaluate the Efficacy and Safety of Racecadotril in Infants, Children and Adolescents With Acute Diarrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RACE3003
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — racecadotril; ORALIT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Racecadotril plus standard treatment oral rehydration solution (Experimental)
  Interventions: Drug: Racecadotril plus ORS
- ORS (standard treatment) (Active Comparator)
  Interventions: Drug: ORS

INTERVENTIONS:
Drug: Racecadotril plus ORS — Racecadotril plus ORS
  Arms: Racecadotril plus standard treatment oral rehydration solution
Drug: ORS — ORS
  Arms: ORS (standard treatment)

SUMMARY:
Multicenter, open-label, controlled, randomized clinical study to evaluate the efficacy and safety of Racecadotril in infants, children and adolescents with acute diarrhea

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from one of the parent(s)/caregiver(s) or subject informed assent
* Children and adolescents, both genders, age from 3 months to < 18 years of age
* Confirmed diagnosis of acute diarrhea (defined as the passage of three or more unformed or liquid stools within the last 24 hours and lasting for less than three days)
* Females of child-bearing potential should agree to continue using a medically acceptable method of birth control throughout the study and for 30 days immediately after the last dose of study drug. Medically acceptable methods of birth control include bilateral tubal ligation or the use of either a contraceptive implant, a contraceptive injection, an intrauterine device, or an oral contraceptive taken within the past three months where the subject agrees to continue using during the study or to adopt another birth control method, or a double-barrier method which consists of a combination of any two of the following: diaphragm, cervical cap, condom, or spermicide

Exclusion Criteria:

* Known allergy to Racecadotril or any of its ingredients
* Subjects suffering from renal or hepatic impairment
* Subjects who need treatment for diarrhea other than ORS alone
* Subjects with fever > 39 degrees Celsius
* Subjects with bloody and/or purulent stools
* Subjects suffering from antibiotic-associated diarrhea, chronic diarrhea or iatrogenic diarrhea
* Subjects with alternating bouts of diarrhea and constipation
* Diarrhea due to exacerbation of chronic gastrointestinal diseases such as irritable bowel syndrome, inflammatory bowel disease or pancreatic exocrine insufficiency
* Cystic fibrosis or coeliac disease
* Subjects suffering from prolonged or uncontrolled vomiting
* Subjects with rare hereditary problems of fructose or galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption syndrome or sucrase isomaltase insufficiency or primary or secondary lactase insufficiency
* Subjects having received antibiotic treatment at any time within 30 days prior to inclusion into the study
* Subjects having received antidiarrheal drugs 48 hours prior to inclusion into the study
* Subjects with severe dehydration required for intravenous/parenteral rehydration
* Subjects who have reported angioedema with angiotensin converting enzyme inhibitors (such as captopril, enalapril, lisinopril, perindopril, ramipril)
* Subjects with combined diseases or medical situations that would prevent to be enrolled depending in the judgment of the investigator
* Intake of experimental drug within 30 days prior to study start
* Subjects with contraindications to ORS or for whom warnings/precautions of ORS apply
* Adolescents (≥ 60 kg) not able to swallow capsules
* Pregnancy and lactation

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Petersburg State Budgetary Healthcare Institution "Municipal Outpatient Children Unit #45", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution | ORS (Standard Treatment)
Started | 62 | 62
Completed | 62 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution | ORS (Standard Treatment) | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 62 | 62 | 124
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.2 (4.5) | 6.8 (4.6) | 6.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 33 | 57
  Male | 38 | 29 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 61 | 59 | 120
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 62 | 62 | 124

OUTCOME MEASURES:

1. Primary Outcome: Duration of Diarrhea (Hours) Between the Start of Treatment Until Last Diarrheal/Watery Stool Before Recovery or End of Study Treatment (Treatment Duration Maximal 5 Days)
Description: Duration of diarrhea is defined by date and time of the evacuation of the final diarrheal stool derived from the daily diary.
  Log-rank test was performed with a p-value < 0.0001
Time Frame: 5 days
Population: full analysis sample
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution | ORS (Standard Treatment)
Number analyzed (Participants) | 62 | 62
hours | 20.0 (2.2) | 43.2 (3.4)

2. Secondary Outcome: Number of Recovered Subjects Per Treatment Group.
Description: Number of recovered subjects per treatment group. Recovery is defined as the evacuation of the first of two consecutive normal stools or no stool within 12 h within treatment period
Time Frame: 5 days
Population: full analysis sample
Measure: Count of Participants; unit: Participants
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution | ORS (Standard Treatment)
Number analyzed (Participants) | 62 | 62
Participants | 62 | 58

3. Secondary Outcome: Number of Recovered Subjects as Defined by Global Physician Assessment of Success at the End of Treatment
Description: Globabl physician assessment used 6 scores with a score of 1 or 2 being regarded as treatment success
Time Frame: 5 days
Population: full analysis sample
Measure: Count of Participants; unit: Participants
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution | ORS (Standard Treatment)
Number analyzed (Participants) | 62 | 62
Participants | 62 | 60

ADVERSE EVENTS:
Time Frame: 5 days + 1 gap day
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution | ORS (Standard Treatment)
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03463512/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03463512/SAP_001.pdf